CLINICAL TRIAL: NCT00789737
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of Welchol as Monotherapy for Type 2 Diabetes Mellitus
Brief Title: Welchol as Monotherapy for Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WEL-305
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Welchol (Experimental): Welchol 625mg tablets
  Interventions: Drug: Welchol
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Welchol — Welchol 625mg tablets
  Arms: Welchol
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
The current study investigates Welchol as monotherapy to improve glycemic control in subjects with Type 2 Diabetes Mellitus not adequately controlled with diet and exercise alone. The study will evaluate if Welchol monotherapy for Type 2 Diabetes Mellitus will be safe, well tolerated and efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >= 18 years of age;
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception as detailed in the protocol.
* Diagnosis of Type 2 Diabetes Mellitus;
* HbA1C >= 7.5% and =< 9.5 % at screening;
* Fasting C-peptide >0.5 ng/mL at screening;
* Drug naïve (no prior treatment with OAD) or having received no pharmacologic therapy for diabetes for the 3 month period prior to screening;
* Clinically stable in regards to medical conditions other than type 2 diabetes;
* Concomitant medications must be at stable doses for at least 30 days prior to enrollment, and are not anticipated to need adjustment during the study period; and
* Fasting glucose =< 240 mg/dL at randomization

Exclusion Criteria:

* A history of type 1 diabetes and/or a history of ketoacidosis;
* History of bowel obstruction;
* History of hypertriglyceridemia-induced pancreatitis;
* Fasting serum triglyceride concentrations >500 mg/dL;
* History of dysphagia, swallowing disorders, gastroparesis, other gastrointestinal (GI) motility disorders, or major GI surgery;
* History of insulin use of >= 2 weeks duration in the previous 3 months or a total of > 2 months of insulin therapy at any time prior to screening;
* Two or more fasting self-monitored blood glucose (SMBG) levels >240 mg/dL during the placebo lead-in period.
* Previous treatment with a bile acid sequestrant, including Welchol within the 3 months prior to screening;
* Body mass index (BMI) >40 kg/m2;
* Weight loss > 3% in prior 3 months; and
* LDL <60 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (90):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Muscle Shoals, Alabama
  - Green Valley, Arizona
  - Mesa, Arizona
  - Tucson, Arizona
  - Searcy, Arkansas
  - Buena Park, California
  - Burbank, California
  - Chula Vista, California
  - Garden Grove, California
  - Huntington Park, California
  - Irvine, California
  - La Mirada, California
  - Lincoln, California
  - Lomita, California
  - Los Angeles, California
  - Los Gatos, California
  - Santa Ana, California
  - Tustin, California
  - Walnut Creek, California
  - Brooksville, Florida
  - Coral Gables, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Gulf Breeze, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Ormond Beach, Florida
  - Pembroke Pines, Florida
  - Vero Beach, Florida
  - Wellington, Florida
  - Winter Park, Florida
  - Decatur, Georgia
  - East Point, Georgia
  - Roswell, Georgia
  - Stockbridge, Georgia
  - Stone Mountain, Georgia
  - Nampa, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - La Porte, Indiana
  - South Bend, Indiana
  - Crestview Hills, Kentucky
  - Lafayette, Louisiana
  - Prince Frederick, Maryland
  - Silver Spring, Maryland
  - New Bedford, Massachusetts
  - Southfield, Michigan
  - Port Gibson, Mississippi
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Clifton, New Jersey
  - Mine Hill, New Jersey
  - New Windsor, New York
  - North Massapequa, New York
  - West Seneca, New York
  - Lexington, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Cuyahoga Falls, Ohio
  - Marion, Ohio
  - Munroe Falls, Ohio
  - Shaker Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Harrisburg, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Arlington, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Manassas, Virginia
  - Salem, Virginia
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Rosenstock J, Rigby SP, Ford DM, Tao B, Chou HS. The glucose and lipid effects of colesevelam as monotherapy in drug-naive type 2 diabetes. Horm Metab Res. 2014 May;46(5):348-53. doi: 10.1055/s-0033-1358759. Epub 2013 Dec 19. PMID 24356792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2009 through July 2011, subjects were recruited from medical clinics, private practice and research clinics.
Pre-assignment Details: There was a 2-week placebo lead-in prior to randomization to treatment arm. Participants were excluded if two or more fasting blood glucose readings >240 mg/dL occurred during lead-in.
  Subjects were excluded if there had been oral antidiabetic, significant insulin, or bile acid sequestrant therapy in the 3 months prior to screening.
Groups:
- Welchol: Welchol 625mg tablets
  Welchol : Welchol 625mg tablets
- Placebo: placebo
  Placebo : placebo
Period: Overall Study
Arm/Group | Welchol | Placebo
Started | 176 | 181
Completed | 128 | 126
Not Completed | 48 | 55
Not completed — Withdrawal by Subject | 13 | 22
Not completed — Lost to Follow-up | 10 | 14
Not completed — Adverse Event | 8 | 8
Not completed — Protocol Violation | 3 | 0
Not completed — Lack of Efficacy | 3 | 0
Not completed — hyperglycemia that met protocol-specifie | 0 | 4
Not completed — Other | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Welchol | Placebo | Total
Number analyzed (Participants) | 176 | 181 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 165 | 167 | 332
  >=65 years | 11 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.25) | 51.8 (10.52) | 52.2 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 92 | 174
  Male | 94 | 89 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 80 | 166
  Not Hispanic or Latino | 90 | 101 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 11 | 23
  Asian | 12 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 29 | 56
  White | 122 | 131 | 253
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 176 | 181 | 357
Body mass index [Mean (Standard Deviation); unit: kg/m*2] | 32.0 (6.5) | 31.8 (4.94) | 31.9 (5.75)
baseline body mass index category [Number; unit: participants] — number >= 30 kg/m*2 and number <30 kg/m*2
  participants
    <30 kg/m*2 | 68 | 66 | 134
    >= 30 kg/m*2 | 108 | 115 | 223
Duration of type 2 diabetes [Mean (Standard Deviation); unit: years] | 4.3 (4.69) | 3.9 (4.39) | 4.1 (4.54)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hemoglobin A1c
Description: change in HbA1c from baseline to Week 24
Time Frame: 24 week
Population: Intent to Treat, Last Observation Carried Forward (LOCF) Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Mean (Standard Error); unit: percentage change of hemoglobin A1c
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 175 | 169
percentage change of hemoglobin A1c | -0.41 (.091) | -0.14 (0.091)
Statistical Analysis 1: Comparison: Welchol vs Placebo; least squares mean; 80% power to detect a 0.3% change; Test type: Superiority or Other; p = 0.0369, ANCOVA

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: to determine changes in Glycemic control after 24 weeks on therapy
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 172 | 166
mg/dL | -4.6 (3.45) [lower limit -19.96] | 5.7 (3.51)
Statistical Analysis 1: Comparison: Welchol vs Placebo; Test type: Superiority or Other; p = 0.0373, ANCOVA

3. Secondary Outcome: % Subjects With a Decrease in HbA1c of >= 0.7 Percentage Units
Description: to determine the percentage of participants who experience a reduction in HbA1c of at least 0.7 percentage units at 24 weeks from baseline.
Time Frame: 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 175 | 169
percentage of participants | 33.1 | 19.5

4. Secondary Outcome: % Subjects Achieving an HbA1C Goal of <7.0
Description: % Subjects achieving an HbA1C goal of <7.0 at 24 weeks
Time Frame: 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 175 | 169
percentage of participants | 20.0 | 13.6

5. Secondary Outcome: % Subjects With a Decrease in FPG >=30 mg/dL
Description: % Subjects with a decrease in Fasting Plasma Glucose >=30 mg/dL from baseline to 24 weeks
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 175 | 169
percentage of participants | 26.9 | 17.8

6. Secondary Outcome: Changes in Total Cholesterol [TC]
Description: To assess the effects of Welchol on changes in total cholesterol [TC]
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 164 | 160
mg/dL | -3.3 (1.02) | 1.8 (1.03)

7. Secondary Outcome: Changes in Low Density Lipoprotein Cholesterol [LDL-C]
Description: To assess the effects of Welchol on changes in low density lipoprotein cholesterol [LDL-C]
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 162 | 160
mg/dL | -10.0 (1.62) | 1.2 (1.63)
Statistical Analysis 1: Comparison: Welchol vs Placebo; Test type: Superiority or Other; p < 0.00001, ANCOVA

8. Secondary Outcome: Changes in High Density Lipoprotein Cholesterol [HDL-C]
Description: To assess the effects of Welchol on changes in high density lipoprotein cholesterol [HDL-C]
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: md/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 164 | 160
md/dL | 1.7 (1.19) | -0.1 (1.21)

9. Secondary Outcome: Changes in Non-HDL-C
Description: To assess the effects of Welchol on changes in non-HDL-C
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 164 | 160
mg/dL | -4.4 (1.34) | 3.0 (1.36)

10. Secondary Outcome: Changes in Triglycerides [TG]
Description: To assess the effects of Welchol on changes in triglycerides [TG]
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 164 | 160
mg/dL | 15.5 (39.82) | 5.8 (38.39)

11. Secondary Outcome: Changes in Apolipoprotein A-I (apoA-I)
Description: To assess the effects of Welchol on changes in apolipoprotein A-I (apoA-I)
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 164 | 160
mg/dL | 3.2 (0.80) | 0.9 (0.81)

12. Secondary Outcome: Changes in Apolipoprotein B (apoB)
Description: To assess the effects of Welchol on changes in apolipoprotein B (apoB)
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 164 | 160
mg/dL | -5.6 (1.18) | 0.9 (1.19)

13. Secondary Outcome: Change in Postprandial Plasma Glucose, 2 Hours After a Meal Tolerance Test
Description: To assess the change from baseline on postprandial plasma glucose, 2 hours after a meal tolerance test
Time Frame: from baseline to 24 weeks
Population: Some participants may not have had lab results for this specific analysis and therefore excluded.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Welchol | Placebo
Number analyzed (Participants) | 131 | 125
mg/dL | -9.3 (5.72) | -1.5 (5.86)

ADVERSE EVENTS:
Time Frame: January 2009 through December 2011
Description: Each visit and phone contact included questions to discover adverse events. The Safety Data Set (Welchol 175 Placebo 171) contains fewer subjects than the Overall Data Set (Welchol 176 Placebo 181) due to the Safety Data Set only includes subjects who took at least 1 dose of study medication and and have at least 1 post-baseline safety measure.
Arm/Group | Welchol | Placebo
Serious Adverse Events (participants affected / at risk) | 7/175 | 3/171
Other Adverse Events (participants affected / at risk) | 91/175 | 77/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Welchol (N=175) | Placebo (N=171)
ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 1 (1)
suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
tibia fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 1 (1) | 1 (1)
psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
coronary artery disease (Vascular disorders) | 2 (2) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
liver function test abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
bilirubin increased (Hepatobiliary disorders) | 1 (2) | 0 (0)
pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Welchol (N=175) | Placebo (N=171)
constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
diarrhoea (Gastrointestinal disorders) | 7 (7) | 3 (3)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1)
bronchitis (Infections and infestations) | 2 (2) | 4 (4)
nasopharyngitis (Infections and infestations) | 2 (2) | 9 (9)
tooth abcess (Infections and infestations) | 4 (4) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2)
urinary tract infection (Infections and infestations) | 7 (7) | 15 (15)
aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2)
blood creatine phosphokinase increased (Investigations) | 4 (4) | 1 (1)
c-reactive protein increased (Investigations) | 6 (6) | 4 (4)
diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
dizziness (Nervous system disorders) | 4 (4) | 4 (4)
headache (Nervous system disorders) | 8 (8) | 5 (5)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
hypertension (Vascular disorders) | 4 (4) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Until coordinated multicenter publication or one year after the study termination, whichever occurs first. After that, submit for Daiichi Sankyo, Inc. (DSI) review and comment at least 45 days before submission. DSI may ask up to 60 additional days, if patentable material is identified.